CLINICAL TRIAL: NCT05661721
Title: Licorice and Home Blood Pressure: a Randomized Crossover Trial
Brief Title: Licorice and Home Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Peder af Geijerstam, Principal investigator, Linkoeping University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: licorice2023
Record Dates: First submitted 2022-12-12; First posted 2022-12-22 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Hypertension,Essential
MeSH Terms: conditions — Essential Hypertension | interventions — Glycyrrhiza glabra extract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention first, control after ("Sweet then salty") (Other): This arm will be divided into the following periods:
  Run-in period: 7 days without any licorice intake Intervention period: 14 days with sweet licorice intake First wash-out period: 14 days without any licorice intake Control period: 14 days with salty licorice intake Second wash-out period: 14 days without any licorice intake.
  Interventions: Other: Sweet licorice; Other: Salty licorice
- Control first, intervention after ("Salty then sweet") (Other): This arm will be divided into the following periods:
  Run-in period: 7 days without any licorice intake Control period: 14 days with salty licorice intake First wash-out period: 14 days without any licorice intake Intervention period: 14 days with sweet licorice intake Second wash-out period: 14 days without any licorice intake.
  Interventions: Other: Sweet licorice; Other: Salty licorice

INTERVENTIONS:
Other: Sweet licorice — Ecologic, vegan and gluten free, low-sodium sweet licorice pastilles made from Glycyrrhiza glabra, with a manufacturer specified content of 4% sugars, 2% glycyrrhizin and 0.03% salt, will be used as intervention. The exact glycyrrhizin content will be determined before the study begins, and participants will be instructed to consume a daily licorice dose that is equivalent to 100 mg of glycyrrhizin.
  Other Names: Glycyrrhiza glabra
Other: Salty licorice — A vegan and gluten free salty licorice without glycyrrhizin, flavored with ammonium chloride, with a manufacturer specified content of 0% sugars and 0.05% salt, will be used as control. The amount of salty licorice will be the same as for sweet licorice, and thus determined after the glycyrrhizin content analysis of the sweet licorice.

SUMMARY:
Out-of-office blood pressure is more strongly associated with cardiovascular risk than office blood pressure. Licorice is known to raise blood pressure, but no previous studies have measured the effects on home blood pressure. The aim of this study is to analyze the association between licorice intake and home blood pressure.

DETAILED DESCRIPTION:
Healthy volunteers will be invited to participate in a randomized, non-blinded, cross-over study. Participants will be randomized to either of two groups with a 1:1 allocation ratio, stratified by sex. Intervention will be sweet licorice and control will be salty licorice. A run-in period of 1 week will be followed by a 2-week intervention/control, a 2-week washout period, another 2-week control/intervention period and again a 2-week washout period. Home blood pressure will be measured continuously, and blood samples (including potassium and aldosterone) will be collected every two weeks. Analyses will be made comparing baseline characteristics of the two groups, intervention/control and washout period results of the two groups to look for potential carry-over effects, and finally comparing intervention and washout period results respectively to the baseline data to look for the effects of licorice.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 30 years

Exclusion Criteria:

* known hypertension, cardiovascular disease, kidney disease, liver disease, hormonal disease, peanut allergy, eating disorder or headache disease (including tension headache and migraine)
* known alcohol abuse or drug abuse (including cannabis and anabolic steroids)
* treatment with hormonal drugs (including oral contraceptives
* known intolerance to licorice intake

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Systolic home blood pressure (mmHg) | Mean at the end of 14 days of intervention compared with mean during run-in period
  Systolic home blood pressure (mmHg)
Diastolic home blood pressure (mmHg) | Mean at the end of 14 days of intervention compared with mean during run-in period
  Diastolic home blood pressure (mmHg)

SECONDARY OUTCOMES:
Body weight (kg) | Mean at the end of 14 days of intervention compared with mean during run-in period
  Body weight (kg)
Plasma potassium (mmol/L) | Mean at the end of 14 days of intervention compared with mean during run-in period
  Plasma potassium (mmol/L)
Plasma sodium (mmol/L) | Mean at the end of 14 days of intervention compared with mean during run-in period
  Plasma sodium (mmol/L)
Plasma renin (mIU/L) | Mean at the end of 14 days of intervention compared with mean during run-in period
  Plasma renin (mIU/L)
Serum aldosterone (μmol/L) | Mean at the end of 14 days of intervention compared with mean during run-in period
  Serum aldosterone (μmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik H Nyström, MD, PhD, Study Director — Linkoeping University
Locations (1):
- Cityhälsan Centrum, Norrköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
As specified below.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After publication in a peer-reviewed journal and for the period of time for which local archive regulations stipulate.
Access Criteria: To be determined on a case by case basis.

REFERENCES:
- [Background] Williams B, Mancia G, Spiering W, Agabiti Rosei E, Azizi M, Burnier M, Clement DL, Coca A, de Simone G, Dominiczak A, Kahan T, Mahfoud F, Redon J, Ruilope L, Zanchetti A, Kerins M, Kjeldsen SE, Kreutz R, Laurent S, Lip GYH, McManus R, Narkiewicz K, Ruschitzka F, Schmieder RE, Shlyakhto E, Tsioufis C, Aboyans V, Desormais I; Authors/Task Force Members:. 2018 ESC/ESH Guidelines for the management of arterial hypertension: The Task Force for the management of arterial hypertension of the European Society of Cardiology and the European Society of Hypertension: The Task Force for the management of arterial hypertension of the European Society of Cardiology and the European Society of Hypertension. J Hypertens. 2018 Oct;36(10):1953-2041. doi: 10.1097/HJH.0000000000001940. PMID 30234752
- [Background] Deutch MR, Grimm D, Wehland M, Infanger M, Kruger M. Bioactive Candy: Effects of Licorice on the Cardiovascular System. Foods. 2019 Oct 14;8(10):495. doi: 10.3390/foods8100495. PMID 31615045
- [Background] Parati G, Stergiou GS, Bilo G, Kollias A, Pengo M, Ochoa JE, Agarwal R, Asayama K, Asmar R, Burnier M, De La Sierra A, Giannattasio C, Gosse P, Head G, Hoshide S, Imai Y, Kario K, Li Y, Manios E, Mant J, McManus RJ, Mengden T, Mihailidou AS, Muntner P, Myers M, Niiranen T, Ntineri A, O'Brien E, Octavio JA, Ohkubo T, Omboni S, Padfield P, Palatini P, Pellegrini D, Postel-Vinay N, Ramirez AJ, Sharman JE, Shennan A, Silva E, Topouchian J, Torlasco C, Wang JG, Weber MA, Whelton PK, White WB, Mancia G; Working Group on Blood Pressure Monitoring and Cardiovascular Variability of the European Society of Hypertension. Home blood pressure monitoring: methodology, clinical relevance and practical application: a 2021 position paper by the Working Group on Blood Pressure Monitoring and Cardiovascular Variability of the European Society of Hypertension. J Hypertens. 2021 Sep 1;39(9):1742-1767. doi: 10.1097/HJH.0000000000002922. PMID 34269334
- [Background] Spinks EA, Fenwick GR. The determination of glycyrrhizin in selected UK liquorice products. Food Addit Contam. 1990 Nov-Dec;7(6):769-78. doi: 10.1080/02652039009373939. PMID 2079112
- [Background] Rizzato G, Scalabrin E, Radaelli M, Capodaglio G, Piccolo O. A new exploration of licorice metabolome. Food Chem. 2017 Apr 15;221:959-968. doi: 10.1016/j.foodchem.2016.11.068. Epub 2016 Nov 17. PMID 27979300
- [Derived] Af Geijerstam P, Joelsson A, Radholm K, Nystrom FH. A low dose of daily licorice intake affects renin, aldosterone, and home blood pressure in a randomized crossover trial. Am J Clin Nutr. 2024 Mar;119(3):682-691. doi: 10.1016/j.ajcnut.2024.01.011. Epub 2024 Jan 20. PMID 38246526